CLINICAL TRIAL: NCT01454245
Title: An Open-Label, Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of JNJ-39439335 Capsule Formulations Administered as a Single Oral Dose in Healthy Male Adult Subjects
Brief Title: A Study to Evaluate the Bioavailability and Food Effect of JNJ-39439335 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR018676; 39439335 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-07-14; First posted 2011-10-18 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: 39439335EDI1013; Bioavailability; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): JNJ-39439335 Part 1:Type=1 unit=mg number=25 form=capsule route=oral use. One capsule (25 mg/day) taken once on Day 1 in 3 treatment periods.
  or Part 1:Type=2 unit=mg number=12.5 form=capsule route=oral use. Two capsules (25 mg/day) taken once on Day 1 in 3 treatment periods.,JNJ-39439335 Part 2:Type=2 unit=mg number=12.5 form=capsule route=oral use. Two capsules taken (25 mg/day) once on Day 1 in 2 treatment periods.
  Interventions: Drug: JNJ-39439335

INTERVENTIONS:
Drug: JNJ-39439335 — Part 2:Type=2, unit=mg, number=12.5, form=capsule, route=oral use. Two capsules taken (25 mg/day) once on Day 1 in 2 treatment periods.
Drug: JNJ-39439335 — Part 1:Type=1, unit=mg, number=25, form=capsule, route=oral use. One capsule (25 mg/day) taken once on Day 1 in 3 treatment periods.
  or Part 1:Type=2, unit=mg, number=12.5, form=capsule, route=oral use. Two capsules (25 mg/day) taken once on Day 1 in 3 treatment periods.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and relative bioavailability of a single dose of 3 capsule formulations of JNJ-39439335 in healthy adult male volunteers. The effect of food on the pharmacokinetics of one of the capsule formulations of JNJ-39439335 will also be evaluated during the study.

DETAILED DESCRIPTION:
This is an open-label (the name of the study drug will be known to the healthy volunteers participating in this study as well as to all study staff), randomized (volunteers will be assigned by chance to 1 of 6 possible treatment sequences of a single dose of 3 different capsule formulations of JNJ-39439335) to evaluate the pharmacokinetics (blood levels of drug) and relative bioavailability (i.e., the rate and extent of absorption of the drug in the body) of JNJ-39439335 (Part 1 of the study). The effect of food on the administration of JNJ-39439335 will then be evaluated on 1 capsule formulation of JNJ-39439335 (Part 2 of the study). The safety and tolerability of JNJ-39439335 will be monitored throughout Part 1 and 2 of the study. In Part 1, healthy volunteers will be randomly assigned to 1 of 6 treatment sequences and will receive a total of 3 single doses of JNJ-39439335. Each dose (2 capsules) will be separated by 21 days. In Part 2, healthy volunteers will be randomly assigned to 1 of 2 treatment sequences and will receive a total of 2 single doses of one formulation selected from Part 1; each dose will be separated by 21 days. Doses will be administered to healthy volunteers under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Have a body mass index (weight [kg]/height2 [m]2) (BMI) between 18 and 30 kg/m2 (inclusive), body weight not less than 50 kg, blood pressure (after sitting for 5 minutes) between 90 and 140 mmHg, systolic, inclusive, and no higher than 90 mmHg diastolic, and an electrocardiogram with results consistent with normal cardiac conduction and function
* Non-smoker for at least 3 months

Exclusion Criteria:

* History of or current medical illness, laboratory values, vital signs, physical examination findings, or electrocardiogram findings deemed clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (Area Under the Curve [AUC]) of JNJ-39439335 | Up to approximately 70 days (14 days after each of 3 doses of study drug in Part I of the study and after each of 2 doses in Part 2 of the study.
Maximum plasma concentration [Cmax]) of JNJ-39439335 | Up to approximately 70 days

SECONDARY OUTCOMES:
No secondary outcome measures are reported

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States